CLINICAL TRIAL: NCT00035659
Title: Longitudinal Study of the Menopause and Fat Patterning
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lynda Powell, PhD, MEd, M.D., Rush University Medical Center
Other Study IDs: 996; R01HL067128 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2015-10

CONDITIONS: Cardiovascular Diseases; Menopause; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To study the natural history of the accumulation of intra-abdominal fat as women progress through the menopause.

DETAILED DESCRIPTION:
BACKGROUND:

Menopause alters the risk for a variety of chronic diseases, including cardiovascular disease, which is the number one cause of mortality in older women. While the associations between menopause, increased total and intra-abdominal fat (IAF), and risk for coronary disease are well established, prospective studies describing the accumulation of IAF, the association with risk factors, and potential mechanistic aspects, are still lacking. This study has the potential to provide important information on the trajectory of IAF accumulation across the menopausal transition in minority and non-minority women.

DESIGN NARRATIVE:

The prospective study will be conducted on an intact biracial cohort of 868 women (419 African Americans; 449 Caucasians) who are participating in a larger study (Women in the Southside Health [WISH] Project) of women undergoing the menopausal transition. This is a population-based cohort that was randomly selected from an existing census with a 72 percent participation rate, approximately equal distribution of socioeconomic status within the African American and Caucasian subgroups, and a dropout rate of only 1 percent/year. As part of the larger study, this cohort undergoes annual exams in which a variety of cardiovascular, hormonal, and lifestyle factors are tracked. These annual measurements consisting of a large number of relevant covariates, including demographics, anthropometrics, serum lipids, blood pressures, insulin, glucose, hormones, lifestyle, health and psychosocial status will be available from the parent study. For this study, two additional clinical tests will be added to the battery at the fourth or fifth annual exam for the 536 women who are expected to be eligible by virtue of not having had a hysterectomy or begun taking hormone therapy. The two tests will be a computed tomography scan for the assessment of intra-abdominal fat, and a dual energy X-ray absorptiometry (DEXA) scan for the assessment of total body fat. These tests will be repeated on an annual basis for the next three years. By the end of the study, it is projected that 462 transitions in menopausal status will have taken place. Random effects models will be used to estimate longitudinal changes in level and rate of intra-abdominal fat as one moves from one menopausal status to another.

ELIGIBILITY:
Women eligible for this ancillary study had no history of diabetes, chronic liver disease or renal disease, no self-reported history of anorexia nervosa, no alcohol or drug abuse, were not currently pregnant or planning to become pregnant, and had not undergone hysterectomy and/or bilateral oophorectomy. Equipment limitations precluded participation of women with breast implants, hip replacements, or weighing ≥299 pounds.

Ages: 42 Years to 61 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The prospective study will be conducted on an intact biracial cohort of 868 women (419 African Americans; 449 Caucasians) who are participating in a larger study (Women in the Southside Health [WISH] Project) of women undergoing the menopausal transition.
Sampling Method: Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2002-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Powell, MD, Principal Investigator — Rush University Medical Center